CLINICAL TRIAL: NCT01993511
Title: Changes in Glucose Metabolism After Roux-en-Y Gastric Bypass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Anna Kirstine Bojsen-Moeller, MD, Hvidovre University Hospital
Other Study IDs: SHJNBJ-FX10
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- RYGB patients with type 2 diabetes: Preoperative oral glucose tolerance test with 2 h P-glucose >11.1 mmol/L
- RYGB patients with IGT: Preoperative oral glucose tolerance test with 2 h p-glucose >7.8 and <11.1 mmol/L
- RYGB patients with NGT: Preoperative oral glucose tolerance test with 2 h p-Glucose <7.8 mmol/L

SUMMARY:
Besides causing weight loss Roux-en-Y gastric bypass (RYGB) has profound effect on glucose metabolism leading to remission of type 2 diabetes early after surgery. However the mechanisms for this improvement remain uncertain. The aim of this study is to investigate the changes in insulin sensitivity and beta-cell function 1 week and 3 months following RYGB using oral and intravenous test.

DETAILED DESCRIPTION:
Investigators plan to study 24 obese patients already enrolled for Roux-en-y gastric bypass surgery (RYGB). 8 with type 2 diabetes (DM2), 8 with impaired glucose tolerance (IGT) and 8 with normal glucose tolerance (NGT) before, within the first week and 3 month after RYGB using a liquid mixed meal test (MMT) and an insulin modified frequently sampled intravenous glucose tolerance test (IM-FSIGT). Furthermore, an oral glucose tolerance test (OGTT) will be performed before and after 3 months. Blood will be sampled in fasting and during the tests measuring plasma glucose, insulin and C-peptid (OGTT, MMT and IM-FSIGT) and GLP-1, glucagon, GIP and GLP-2 (MMT). Beta-cell function will be assessed from the MMT (insulinogenic index - IGI), OGTT (IGI) and the IM-FSIGT (Acute insulin response, AIR) in order to examine whether changes in beta-cell function after RYGB depend on an oral stimulus. Insulin sensitivity will be assessed in fasting (HOMA-IR), during the IM-FSIGT (minimal model: Si) and from MMT/OGTT (Matsuda index). Insulin clearance/hepatic extraction of insulin will be assessed in fasting and during the intravenous and oral test.

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for RYGB, Age 18-60 years, BMI 35-60 kg/m2 at time of referral to operation, blood pressure <145/85, C-peptid>700 pmol/l.

Exclusion Criteria:

* Obesity caused by medical treatment for psychiatric disease. Mental retardation. Alcohol or drug abuse. Severe cardiopulmonary disease. History of peritonitis, ventricular disease, upper gastrointestinal surgery, recurrent oesophagitis or severe complications to general anesthesia. Bad compliance. Treatment with thyroid hormones or antithyroid treatment. Treatment with anorectic medicine later than 3 months prior to surgery. Furthermore prior to surgery each patient has to loose 8 % of bodyweight to reduce the risk of operative complications.

Before each test day all glucose lowering medication will be paused for an appropriate amount of time depending on the type of medicine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Morbid obese patients who are already enrolled for Roux-en-y gastric bypass surgery will be invited to participate (investigators do not assign patients to the surgery). 8 with type 2 diabetes, 8 with impaired glucose tolerance and 8 with normal glucose tolerance. Glucose tolerance will be assessed with an oral glucose tolerance test (OGTT) prior to surgery and prior to the other tests. Plasma glucose 120 minutes after OGTT will define glucose tolerance. Normal: < 7,8 mM. Impaired: 7,8 - 11,1 mM. Diabetic: >11,1 mM.
  Subjects are recruited from the outpatient clinic of endocrinology and gastrosurgical clinic at Hvidovre University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change in beta-cell function after RYGB. | 1 week and 3 months.
  Beta-cell function will be assessed with both intravenous tests (acute insulin response to glucose - AIRg) and oral tests (insulinogenic index - IGI).

SECONDARY OUTCOMES:
Change in insulin sensitivity after RYGB. | 1 week and 3 months.
  Insulin sensitivity will be assessed in fasting and by intravenous tests (sensitivity index - Si) and oral tests (Matsuda index).

OTHER OUTCOMES:
Change in glucagon and gastrointestinal hormone secretion after RYGB. | 1 week and 3 months
Change in insulin clearance after RYGB. | 1 week and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kirstine Bojsen-Moeller, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Palleja A, Kashani A, Allin KH, Nielsen T, Zhang C, Li Y, Brach T, Liang S, Feng Q, Jorgensen NB, Bojsen-Moller KN, Dirksen C, Burgdorf KS, Holst JJ, Madsbad S, Wang J, Pedersen O, Hansen T, Arumugam M. Roux-en-Y gastric bypass surgery of morbidly obese patients induces swift and persistent changes of the individual gut microbiota. Genome Med. 2016 Jun 15;8(1):67. doi: 10.1186/s13073-016-0312-1. PMID 27306058
- [Derived] Martinussen C, Bojsen-Moller KN, Dirksen C, Jacobsen SH, Jorgensen NB, Kristiansen VB, Holst JJ, Madsbad S. Immediate enhancement of first-phase insulin secretion and unchanged glucose effectiveness in patients with type 2 diabetes after Roux-en-Y gastric bypass. Am J Physiol Endocrinol Metab. 2015 Mar 15;308(6):E535-44. doi: 10.1152/ajpendo.00506.2014. Epub 2015 Jan 27. PMID 25628424